CLINICAL TRIAL: NCT06170242
Title: A Randomized, Phase 2a, Double-blind, Placebo-controlled Study to Evaluate the Safety, Pharmacokinetics and Antiviral Activity of Multiple Doses of Orally Administered EDP-323 Against Respiratory Syncytial Virus Infection in a Virus Challenge Model in Healthy Adults
Brief Title: A Controlled Phase 2a Study to Evaluate the Efficacy of EDP-323 Against Respiratory Syncytial Virus Infection in a Virus Challenge Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: hVIVO Services Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDP 323-101
Record Dates: First submitted 2023-11-27; First posted 2023-12-14 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: RSV Infection
Keywords: challenge study; RSV; antiviral; RSV-A Memphis 37b
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EDP-323 Arm A (Experimental): Subjects will take EDP-323 Dose 1 orally for 5 days
  Interventions: Drug: EDP-323 Dose Regimen 1
- EDP-323 Arm B (Experimental): Subjects will take EDP-323 Dose 2 orally for 5 days
  Interventions: Drug: EDP-323 Dose Regimen 2
- Placebo Arm C (Placebo Comparator): Subjects will take matching placebo orally for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-323 Dose Regimen 1 — EDP-323 capsule
  Arms: EDP-323 Arm A
Drug: EDP-323 Dose Regimen 2 — EDP-323 capsule
  Arms: EDP-323 Arm B
Drug: Placebo — Placebo capsule
  Arms: Placebo Arm C

SUMMARY:
A randomized, Phase 2a, double-blind, placebo-controlled study to evaluate the safety, pharmacokinetics and antiviral activity of multiple doses of orally administered EDP-323 in healthy subjects infected with RSV-A Memphis 37b. This study is designed to assess the antiviral effect of EDP-323 compared to a placebo control in the respiratory syncytial virus challenge model.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Age 18 to 55 years, inclusive.
* In good health with no history of major medical conditions.
* A total body weight ≥ 50 kg and Body Mass Index (BMI) ≥ 18 kg/m2 and ≤ 35kg/m2.

Exclusion Criteria:

* Pregnant or nursing females
* Acute or chronic medical illness
* History of, or currently active, symptoms or signs suggestive of upper or lower respiratory tract (URT or LRT) infection within 4 weeks prior to the first study visit.
* Abnormal lung function
* Positive for HIV, active hepatitis B or C test
* Nose or nasopharynx abnormalities
* Receipt of any investigational drug within 3 months prior to the planned date of viral challenge/first dose of study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- hVIVO Services Limited, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 142 participants were enrolled and inoculated with challenge virus (Respiratory Syncytial Virus [RSV]-A Memphis 37b) of which 141 participants were randomized 1:1:1 into one of three treatment groups to receive EDP-323 (at two different doses) or placebo at one site in the United Kingdom between November 2023 and July 2024.
Pre-assignment Details: One participant was enrolled and received RSV-A Memphis 37b virus inoculation on Day 0 but was not randomized to receive EDP-323 or matched placebo.
Groups:
- EDP-323 High Dose: Participants received RSV-A Memphis 37b virus inoculation on Day 0 then orally administered 600 mg EDP-323 once daily (QD) for 5 days.
- EDP-323 Low Dose: Participants received RSV-A Memphis 37b virus inoculation on Day 0 then orally administered loading dose 600 mg EDP-323 on Day 1 followed by 200 mg EDP-323 QD for the remaining 4 days.
- Placebo: Participants received RSV-A Memphis 37b virus inoculation on Day 0 then orally administered matching placebo QD for 5 days.
- Enrolled But Not Randomized: Participant received RSV-A Memphis 37b virus inoculation on Day 0 but was not randomized to receive EDP-323 or matched placebo.
Period: Overall Study
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo | Enrolled But Not Randomized
Started | 47 | 47 | 47 | 1
Completed | 47 | 47 | 46 | 0
Not Completed | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (Treated Participants): All participants having received challenge virus and investigational medicinal product (IMP).
Groups:
- EDP-323 High Dose: Participants received RSV-A Memphis 37b virus inoculation on Day 0 then orally administered 600 mg EDP-323 QD for 5 days.
- Total: Total of all reporting groups
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo | Total
Number analyzed (Participants) | 47 | 47 | 47 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.09 (6.372) | 27.62 (5.980) | 27.91 (6.223) | 28.21 (6.182)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 19 | 51
  Male | 32 | 30 | 28 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 39 | 35 | 38 | 112
  Black or African American | 3 | 7 | 5 | 15
  Asian | 2 | 3 | 1 | 6
  Other | 3 | 2 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 46 | 45 | 46 | 137

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Reverse Transcription-polymerase Chain Reaction (qRT-PCR): RSV Area Under the Viral Load-time Curve (VL-AUC)
Description: Measured by qRT-PCR in nasal samples.
Time Frame: Day 1 to Day 12
Population: Intent-to-treat infected (ITT-I) Analysis Set: All participants having received challenge virus, randomized, and having received at least one dose of IMP, and meeting the criterion for laboratory-confirmed RSV infection.
Measure: Mean (Standard Deviation); unit: log10 copies/mL*hours
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 26 | 23 | 30
log10 copies/mL*hours | 99.05 (133.325) | 82.28 (158.033) | 657.45 (396.743)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose versus (vs) Placebo; Test type: Superiority — P-values are from analysis of covariance (ANCOVA) with treatment group as main effect and the baseline value as a covariate. The baseline value is defined as the qRT-PCR viral load value at the time of first dose of IMP; p < 0.0001, ANCOVA; Difference in least square (LS) means = -540.56, 95% CI 2-sided [-680.80 to -400.33]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Low Dose vs Placebo; Test type: Superiority — P-values are from ANCOVA with treatment group as main effect and the baseline value as a covariate. The baseline value is defined as the qRT-PCR viral load value at the time of first dose of IMP; p < 0.0001, ANCOVA; Difference in LS mean = -523.12, 95% CI 2-sided [-674.46 to -371.78]
Statistical Analysis 3: Comparison: EDP-323 High Dose vs EDP-323 Low Dose vs Placebo; Pooled EDP-323 vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, ANCOVA; Difference in LS means = -536.30, 95% CI 2-sided [-641.71 to -430.89]

2. Secondary Outcome: qRT-PCR: RSV Peak Viral Load (VLPEAK)
Description: Measured by qRT-PCR in nasal samples.
Time Frame: Day 1 to Day 12
Population: ITT-I Analysis Set: All participants having received challenge virus, randomized, and having received at least one dose of IMP, and meeting the criterion for laboratory-confirmed RSV infection.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 26 | 23 | 30
log10 copies/mL | 2.52 (2.173) | 1.99 (2.711) | 6.48 (2.311)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, ANCOVA; Difference in LS mean = -3.83, 95% CI 2-sided [-4.85 to -2.81]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Low Dose vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, ANCOVA; Difference in LS mean = -4.16, 95% CI 2-sided [-5.44 to -2.89]

3. Secondary Outcome: qRT-PCR: Time From the Assessment at the Time of the First Dose of IMP to RSV VLPEAK
Description: Measured by qRT-PCR in nasal samples.
Time Frame: Day 1 to Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 26 | 23 | 30
days | 2.89 (2.922) | 3.12 (3.113) | 3.12 (1.555)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.6330, ANCOVA; Difference in LS mean = -0.29, 95% CI 2-sided [-1.50 to 0.92]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Lose Dose vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.8309, ANCOVA; Difference in LS mean = -0.14, 95% CI 2-sided [-1.46 to 1.17]

4. Secondary Outcome: qRT-PCR: Time From the Assessment at the Time of the First Dose of IMP to RSV Viral Load Negativity
Description: The time from the assessment at the time of the first dose of IMP to qRT-viral load negativity was analyzed using the Kaplan-Meier method. Viral load negativity was reached at the first time when the viral load was undetectable (< lower limit of detection [LLOD]) by qRT-PCR, after which no further detectable assessment appeared. Measured by qRT-PCR in nasal samples.
Time Frame: Day 1 to Day 12
Population: ITT-I Analysis Set: All participants having received challenge virus, randomized, and having received at least one dose of IMP, and meeting the criterion for laboratory-confirmed RSV infection. Inclusive only of participants with available data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 20 | 17 | 30
days | 2.3 [1.0 to 6.5] | 1.5 [0.5 to 6.0] | 8.5 [6.5 to NA] — Upper confidence interval was not reached due to lack of events and the upper bound extending beyond the largest observed time for this group.

5. Secondary Outcome: qRT-PCR: Time From the Assessment at the Time of the First Dose of IMP to First Negative Slope of RSV Viral Load
Description: Time to first negative slope = time of the timepoint after which there are two consecutive declines in viral load - time of the nearest viral load assessment to the first dose of IMP. Measured by qRT-PCR in nasal samples.
Time Frame: Day 1 to Day 12
Population: ITT-I Analysis Set: All participants having received challenge virus, randomized, and having received at least one dose of IMP, and meeting the criterion for laboratory-confirmed RSV infection. Inclusive only of participants with at least one detectable viral load during qRT-PCR.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 13 | 9 | 27
days | 0.77 (0.954) | 1.33 (2.360) | 2.60 (1.632)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.0021, ANCOVA; Difference in LS mean = -1.57, 95% CI 2-sided [-2.53 to -0.61]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Lose Dose vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.0905, ANCOVA; Difference in LS mean = -1.09, 95% CI 2-sided [-2.35 to 0.18]

6. Secondary Outcome: qRT-PCR: RSV Viral Load Clearance Rate - EDP-323 High Dose
Description: Calculated as the slope of the RSV viral load over time from time of RSV VLPEAK to 1, 2, 3, and 4 days later. Estimates for fixed effects of a mixed linear model, modeling the viral load from peak up to the 4 following days, with time from VLPEAK, group and interaction between time and group as fixed effects and a random intercept within each participant. The model was a distinct analysis for the EDP-323 high dose and placebo groups where the estimates for both groups are model-dependent and impacted by the overall model. A negative slope indicated that the viral load decreased over time. Measured by qRT-PCR in nasal samples.
Time Frame: Up to Day 16
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: log10 copies/mL/day
Arm/Group | EDP-323 High Dose | Placebo
Number analyzed (Participants) | 17 | 28
log10 copies/mL/day | -0.5650 [-0.7539 to -0.3761] | -1.3299 [-1.4775 to -1.1823]

7. Secondary Outcome: qRT-PCR: RSV Viral Load Clearance Rate - EDP-323 Low Dose
Description: Calculated as the slope of the RSV viral load over time from time of RSV VLPEAK to 1, 2, 3, and 4 days later. Estimates for fixed effects of a mixed linear model, modeling the viral load from peak up to the 4 following days, with time from VLPEAK, group and interaction between time and group as fixed effects and a random intercept within each participant. The model was a distinct analysis for the EDP-323 low dose and placebo groups where the estimates for both groups are model-dependent and impacted by the overall model. A negative slope indicated that the viral load decreased over time. Measured by qRT-PCR in nasal samples.
Time Frame: Up to Day 16
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: log10 copies/mL/day
Arm/Group | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 10 | 28
log10 copies/mL/day | -0.5480 [-0.8182 to -0.2778] | -1.3298 [-1.4896 to -1.1699]

8. Secondary Outcome: Viral Culture: RSV VL-AUC
Description: Measured by viral culture (plaque assay) in nasal samples.
Time Frame: Day 1 to Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 plaque-forming units (PFU)/mL*h
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 26 | 23 | 30
log10 plaque-forming units (PFU)/mL*h | 3.82 (9.333) | 6.21 (15.448) | 227.04 (189.998)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — P-values are from ANCOVA with treatment group as main effect and the baseline value as a covariate. The baseline value is defined as the cell culture viral load value at the time of first dose of IMP; p < 0.0001, ANCOVA; Difference in LS mean = -203.63, 95% CI 2-sided [-272.18 to -135.07]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Low Dose vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.0001, ANCOVA; Difference in LS mean = -215.03, 95% CI 2-sided [-288.84 to -141.22]

9. Secondary Outcome: Viral Culture: RSV VLPEAK
Description: Measured by viral culture (plaque assay) in nasal samples.
Time Frame: Day 1 to Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 PFU/mL
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 26 | 23 | 30
log10 PFU/mL | 0.04 (0.198) | 0.16 (0.569) | 3.45 (2.191)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.0001, ANCOVA; Difference in LS mean = -3.22, 95% CI 2-sided [-4.05 to -2.40]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Low Dose vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.0001, ANCOVA; Difference in LS mean = -3.23, 95% CI 2-sided [-4.11 to -2.34]

10. Secondary Outcome: Viral Culture: Time From the Assessment at the Time of the First Dose of IMP to RSV VLPEAK
Description: Measured by viral culture (plaque assay) in nasal samples.
Time Frame: Day 1 to Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 26 | 23 | 30
days | 5.82 (2.980) | 5.78 (3.304) | 3.95 (2.290)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0238, ANCOVA; Difference in LS mean = 1.44, 95% CI 2-sided [0.20 to 2.68]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Low Dose vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0134, ANCOVA; Difference in LS mean = 1.68, 95% CI 2-sided [0.36 to 2.99]

11. Secondary Outcome: Viral Culture: Time From the Assessment at the Time of the First Dose of IMP to RSV Viral Load Negativity
Description: Measured by viral culture (plaque assay) in nasal samples.
Time Frame: Day 1 to Day 12
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 6 | 6 | 23
days | 0.5 [0.5 to NA] — Upper confidence interval was not reached due to lack of events. | 0.5 [0.5 to NA] — Upper confidence interval was not reached due to lack of events. | 4.5 [4.5 to 5.5]

12. Secondary Outcome: Viral Culture: Time From the Assessment at the Time of the First Dose of IMP to First Negative Slope of RSV Viral Load
Description: Measured by viral culture (plaque assay) in nasal samples.
Time Frame: Day 1 to Day 12
Population: ITT-I Analysis Set: All participants having received challenge virus, randomized, and having received at least one dose of IMP, and meeting the criterion for laboratory-confirmed RSV infection. Inclusive only of participants with at least one detectable viral load during plaque assay.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 3 | 3 | 23
days | 0.00 (0.000) | 0.00 (0.000) | 2.92 (1.739)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0389, ANCOVA; Difference in LS mean = -2.18, 95% CI 2-sided [-4.23 to -0.12]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Low Dose vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.2713, ANCOVA; Difference in LS mean = -1.31, 95% CI 2-sided [-3.73 to 1.10]

13. Secondary Outcome: Viral Culture: RSV Viral Load Clearance Rate
Description: Calculated as the slope of the RSV viral load over time from time of RSV VLPEAK to 1, 2, 3, and 4 days later. Estimates for fixed effects of a mixed linear model, modeling the viral load from peak up to the 4 following days, with time from VLPEAK, group and interaction between time and group as fixed effects and a random intercept within each participant. A negative slope indicated that the viral load decreased over time. Measured by viral culture in nasal samples.
Time Frame: Up to Day 16
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: log10 PFU/mL/day
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 3 | 3 | 23
log10 PFU/mL/day | -0.1336 [-0.7642 to 0.4970] | -0.2565 [-0.6990 to 0.1861] | -1.1124 [-1.2522 to -0.9727]

14. Secondary Outcome: Area Under the Total Symptom Score (TSS)-Time Curve (TSS-AUC)
Description: An individual TSS (10-items) was derived at each assessment of the diary card as the sum of the scores given to the 10 following symptoms on that symptom score card, giving a score between 0 and 3:
  * Runny nose
  * Stuffy nose
  * Sneezing
  * Sore throat
  * Earache
  * Malaise/Tiredness
  * Headache
  * Muscle and/or Joint Ache
  * Cough
  * Shortness of breath
  TSS ranged from 0 to 30 with higher TSS indicating a higher disease burden and thus a worse outcome.
  The calculation of the TSS-AUC was performed on the TSS measured 3 times a day using the trapezoidal summation rule based on actual time intervals in hours.
Time Frame: Day 1 to Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score*hours
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 26 | 23 | 30
score*hours | 127.31 (149.221) | 82.67 (100.412) | 369.10 (330.397)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — P-values are from ANCOVA with treatment group as main effect and the baseline value as a covariate. The baseline value is defined as the TSS value at the time of first dose of IMP; p < 0.0001, ANCOVA; Difference in LS mean = -280.61, 95% CI 2-sided [-404.44 to -156.77]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Low Dose vs Placebo; Test type: Superiority — [test comment as in outcome 14, analysis 1]; p < 0.0001, ANCOVA; Difference in LS mean = -301.15, 95% CI 2-sided [-428.53 to -173.76]

15. Secondary Outcome: Peak TSS
Description: Defined as the highest recorded value of TSS.
  An individual TSS (10-items) was derived at each assessment of the diary card as the sum of the scores given to the 10 following symptoms on that symptom score card, giving a score between 0 and 3:
  * Runny nose
  * Stuffy nose
  * Sneezing
  * Sore throat
  * Earache
  * Malaise/Tiredness
  * Headache
  * Muscle and/or Joint Ache
  * Cough
  * Shortness of breath
  TSS ranged from 0 to 30 with higher TSS indicating a higher disease burden and thus a worse outcome.
Time Frame: Day 1 to Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 26 | 23 | 30
score on a scale | 2.65 (1.765) | 2.35 (2.673) | 5.77 (4.439)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — [test comment as in outcome 14, analysis 1]; p < 0.0001, ANCOVA; Difference in LS mean = -3.64, 95% CI 2-sided [-5.26 to -2.02]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Low Dose vs Placebo; Test type: Superiority — [test comment as in outcome 14, analysis 1]; p < 0.0001, ANCOVA; Difference in LS mean = -3.70, 95% CI 2-sided [-5.35 to -2.05]

16. Secondary Outcome: Time to Peak TSS
Description: Time to peak TSS = time of peak TSS - time of the nearest TSS assessment to the first dose of IMP.
  An individual TSS (10-items) was derived at each assessment of the diary card as the sum of the scores given to the 10 following symptoms on that symptom score card, giving a score between 0 and 3:
  * Runny nose
  * Stuffy nose
  * Sneezing
  * Sore throat
  * Earache
  * Malaise/Tiredness
  * Headache
  * Muscle and/or Joint Ache
  * Cough
  * Shortness of breath
  TSS ranged from 0 to 30 with higher TSS indicating a higher disease burden and thus a worse outcome.
Time Frame: Day 1 to Day 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 26 | 23 | 30
days | 2.00 (2.403) | 2.84 (3.125) | 3.36 (2.065)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — [test comment as in outcome 14, analysis 1]; p = 0.0552, ANCOVA; Difference in LS mean = -1.08, 95% CI 2-sided [-2.19 to 0.03]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Low Dose vs Placebo; Test type: Superiority — [test comment as in outcome 14, analysis 1]; p = 0.5599, ANCOVA; Difference in LS mean = -0.38, 95% CI 2-sided [-1.69 to 0.92]

17. Secondary Outcome: Time to Resolution From Peak TSS
Description: Time to resolution from peak TSS = time of the first 24-hour symptom-free time point - time of peak TSS.
  An individual TSS (10-items) was derived at each assessment of the diary card as the sum of the scores given to the 10 following symptoms on that symptom score card, giving a score between 0 and 3:
  * Runny nose
  * Stuffy nose
  * Sneezing
  * Sore throat
  * Earache
  * Malaise/Tiredness
  * Headache
  * Muscle and/or Joint Ache
  * Cough
  * Shortness of breath
  TSS ranged from 0 to 30 with higher TSS indicating a higher disease burden and thus a worse outcome.
Time Frame: Day 1 to Day 12
Population: ITT-I Analysis Set: All participants having received challenge virus, randomized, and having received at least one dose of IMP, and meeting the criterion for laboratory-confirmed RSV infection. Inclusive of participants with at least one TSS >0 only.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 24 | 16 | 28
days | 2.16 (1.922) | 2.58 (2.415) | 2.93 (1.789)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — [test comment as in outcome 14, analysis 1]; p = 0.0307, ANCOVA; Difference in LS mean = -1.04, 95% CI 2-sided [-1.97 to -0.10]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Test type: Superiority — [test comment as in outcome 14, analysis 1]; p = 0.4119, ANCOVA; Difference in LS mean = -0.53, 95% CI 2-sided [-1.81 to 0.76]

18. Secondary Outcome: Total Weight of Nasal Discharge (Mucus) Produced
Description: Each participant was given pre-weighed packets of paper tissues. Participants were asked to place single tissues used for nose blowing or sneezing into a specified collection bag (for that participant only).
Time Frame: Day 1 to Day 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 26 | 23 | 29
grams | 6.12 (6.564) | 9.49 (20.537) | 16.44 (22.152)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — P-values are from ANCOVA with treatment group as main effect and the baseline value as a covariate. The baseline value is defined as the biospecimen value at the time of first dose of IMP; p = 0.0042, ANCOVA; Difference in LS mean = -13.37, 95% CI 2-sided [-22.34 to -4.40]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Low Dose vs Placebo; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.0058, ANCOVA; Difference in LS mean = -13.19, 95% CI 2-sided [-22.38 to -4.00]

19. Secondary Outcome: Total Number of Tissues Used
Description: as for outcome 18
Time Frame: Day 1 to Day 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: tissues
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 26 | 23 | 29
tissues | 17.62 (23.329) | 16.22 (21.457) | 28.79 (27.580)
Statistical Analysis 1: Comparison: EDP-323 High Dose vs Placebo; High Dose vs Placebo; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.0026, ANCOVA; Difference in LS mean = -18.72, 95% CI 2-sided [-30.61 to -6.84]
Statistical Analysis 2: Comparison: EDP-323 Low Dose vs Placebo; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p = 0.0022, ANCOVA; Difference in LS mean = -19.28, 95% CI 2-sided [-31.30 to -7.26]

20. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Plasma pharmacokinetic (PK) parameters for EDP-323 and metabolites (EP-038725 and EP-039082) were estimated using non-compartmental methods. The plasma PK parameters were estimated from the concentration-time profiles. In estimating the PK parameters, below the limit of quantification (BQL) values were set to zero. Actual sampling times, rather than scheduled sampling times, were used in all computations involving sampling times. If the actual time or dose time was missing, the scheduled time could be substituted in order to calculate the PK parameter.
  In case of an actual sampling time deviating by >20% from the scheduled (nominal) time, this plasma concentration was excluded from descriptive statistics in the plasma concentration-time table.
Time Frame: First Dose: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, and 15 hours post-dose) and Day 2 pre-dose; Last Dose: Day 5 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, 48, 60, and 72 hours post-dose)
Population: PK Analysis Set: All ITT analysis set participants with at least one post-dose PK result. Inclusive only of participants with available data for each analyte and timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose
Number analyzed (Participants) | 47 | 47
ng/mL
  First Dose: EDP-323 | 1358.47 (590.191) | 1453.70 (627.552)
  Last Dose: EDP-323 | 1703.09 (746.730) | 759.38 (322.938)
  First Dose: EP-038725 | 1225.02 (753.882) | 1501.55 (776.020)
  Last Dose: EP-038725 | 1294.19 (772.921) | 381.94 (266.839)
  First Dose: EP-039082 | 5.40 (5.265) | 6.59 (4.923)
  Last Dose: EP-039082 | 6.41 (5.131) | 1.40 (1.346)

21. Secondary Outcome: Time to Cmax (Tmax)
Description: Plasma PK parameters for EDP-323 and metabolites (EP-038725 and EP-039082) were estimated using non-compartmental methods. The plasma PK parameters were estimated from the concentration-time profiles. In estimating the PK parameters, BQL values were set to zero. Actual sampling times, rather than scheduled sampling times, were used in all computations involving sampling times. If the actual time or dose time was missing, the scheduled time could be substituted in order to calculate the PK parameter.
  In case of an actual sampling time deviating by >20% from the scheduled (nominal) time, this plasma concentration was excluded from descriptive statistics in the plasma concentration-time table.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose
Number analyzed (Participants) | 47 | 47
hours
  First Dose: EDP-323 | 3.98 [1.0 to 10.2] | 3.92 [1.9 to 9.9]
  Last Dose: EDP-323 | 4.82 [2.0 to 9.9] | 4.10 [1.0 to 10.3]
  First Dose: EP-038725 | 3.97 [1.9 to 10.2] | 3.85 [1.9 to 9.9]
  Last Dose: EP-038725 | 4.92 [2.0 to 9.9] | 3.98 [1.0 to 10.0]
  First Dose: EP-039082 | 3.00 [0.0 to 9.9] | 2.97 [0.9 to 9.9]
  Last Dose: EP-039082 | 3.82 [1.0 to 9.9] | 2.00 [0.0 to 7.9]

22. Secondary Outcome: Terminal Half-life (t1/2)
Description: as for outcome 21
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, and 15 hours post-dose), Day 2 pre-dose, Day 3 pre-dose, Day 4 pre-dose, Day 5 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, 48, 60, and 72 hours post-dose)
Population: PK Analysis Set: All ITT analysis set participants with at least one post-dose PK result. Inclusive only of participants with available data for each analyte and timepoint. No participants in the EDP-323 low dose group had quantifiable samples for EP-039082 (below limit of quantification [BLQ]) for the analysis of this PK parameter.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose
Number analyzed (Participants) | 46 | 46
hours
  EDP-323 | 13.07 (4.793) | 12.55 (4.621)
  EP-038725: number analyzed (Participants) | 33 | 37
  EP-038725 | 16.56 (3.049) | 17.16 (3.103)
  EP-039082: number analyzed (Participants) | 3 | 0
  EP-039082 | 3.89 (1.346) |

23. Secondary Outcome: Apparent Systemic Clearance at Steady-state (CLss/F)
Description: as for outcome 21
Time Frame: as for outcome 22
Population: PK Analysis Set: All ITT analysis set participants with at least one post-dose PK result. Inclusive only of participants with available data for each analyte and timepoint. No participants in the EDP-323 high dose and EDP-323 low dose groups had quantifiable samples for EP-038725 and EP-039082 (BLQ) for the analysis of this PK parameter.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose
Number analyzed (Participants) | 46 | 46
L/h
  EDP-323 | 32.39 (13.648) | 24.51 (11.383)
  EP-038725: number analyzed (Participants) | 0 | 0
  EP-039082: number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Terminal Elimination Rate Constant (λz)
Description: as for outcome 21
Time Frame: as for outcome 22
Population: PK Analysis Set: All ITT analysis set participants with at least one post-dose PK result. Inclusive only of participants with available data for each analyte and timepoint. No participants in the EDP-323 low dose group had quantifiable samples for EP-039082 (BLQ) for the analysis of this PK parameter.
Measure: Mean (Standard Deviation); unit: per hour
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose
Number analyzed (Participants) | 46 | 46
per hour
  EDP-323 | 0.06 (0.018) | 0.06 (0.019)
  EP-038725: number analyzed (Participants) | 33 | 37
  EP-038725 | 0.04 (0.009) | 0.04 (0.008)
  EP-039082: number analyzed (Participants) | 6 | 0
  EP-039082 | 0.17 (0.061) |

25. Secondary Outcome: Apparent Volume of Distribution at Steady-state (Vss/F)
Description: as for outcome 21
Time Frame: as for outcome 22
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose
Number analyzed (Participants) | 46 | 46
liters
  EDP-323 | 569.26 (208.202) | 402.73 (143.305)
  EP-038725: number analyzed (Participants) | 0 | 0
  EP-039082: number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Plasma Concentration at 12 Hours (C12h) and 24 Hours (C24h)
Description: In case of an actual sampling time deviating by >20% from the scheduled (nominal) time, this plasma concentration was excluded from descriptive statistics in the plasma concentration-time table.
Time Frame: First Dose: Day 1, 12 and 24 hours post-dose; Last Dose: Day 5, 12 and 24 hours post-dose
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose
Number analyzed (Participants) | 47 | 47
ng/mL
  First Dose C12h: EDP-323 | 711.96 (265.557) | 756.02 (345.633)
  First Dose C24h: EDP-323: number analyzed (Participants) | 46 | 46
  First Dose C24h: EDP-323 | 351.45 (166.086) | 368.54 (216.140)
  Last Dose C12h: EDP-323 | 935.04 (318.005) | 423.38 (203.294)
  Last Dose C24h: EDP-323 | 493.16 (250.229) | 220.69 (141.715)
  First Dose C12h: EP-038725 | 189.71 (94.962) | 221.48 (162.256)
  First Dose C24h: EP-038725: number analyzed (Participants) | 46 | 46
  First Dose C24h: EP-038725 | 52.47 (27.362) | 56.57 (23.845)
  Last Dose C12h: EP-038725 | 281.01 (168.564) | 78.22 (39.056)
  Last Dose C24h: EP-038725 | 96.78 (59.546) | 30.29 (14.620)
  First Dose C12h: EP-039082 | 1.28 (0.493) | 1.44 (0.775)
  First Dose C24h: EP-039082: number analyzed (Participants) | 46 | 46
  First Dose C24h: EP-039082 | 1.00 (0.000) | 1.01 (0.041)
  Last Dose C12h: EP-039082 | 1.60 (0.739) | 1.00 (0.014)
  Last Dose C24h: EP-039082 | 1.04 (0.166) | 1.00 (0.000)

27. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration (AUC0-last)
Description: Plasma PK parameters for EDP-323 and metabolites (EP-038725 and EP-039082) were estimated using non-compartmental methods. The AUCs were calculated using linear up/log down method. In estimating the PK parameters, BQL values were set to zero. Actual sampling times, rather than scheduled sampling times, were used in all computations involving sampling times. If the actual time or dose time was missing, the scheduled time could be substituted in order to calculate the PK parameter.
  In case of an actual sampling time deviating by >20% from the scheduled (nominal) time, this plasma concentration was excluded from descriptive statistics in the plasma concentration-time table.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose
Number analyzed (Participants) | 47 | 47
h*ng/mL
  First Dose: EDP-323 | 15626.46 (5982.746) | 16703.77 (7268.939)
  Last Dose: EDP-323 | 31084.37 (13945.732) | 13816.76 (7801.297)
  First Dose: EP-038725 | 7181.42 (3848.438) | 8319.19 (3563.734)
  Last Dose: EP-038725 | 10814.63 (5619.005) | 3174.73 (1641.754)
  First Dose: EP-039082: number analyzed (Participants) | 43 | 47
  First Dose: EP-039082 | 26.11 (21.928) | 31.34 (28.251)
  Last Dose: EP-039082: number analyzed (Participants) | 47 | 33
  Last Dose: EP-039082 | 35.35 (28.171) | 4.77 (4.119)

28. Secondary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUC0-tau)
Description: as for outcome 27
Time Frame: Last Dose: Day 5 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, 48, 60, and 72 hours post-dose)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose
Number analyzed (Participants) | 47 | 47
h*ng/mL
  Last Dose: EDP-323 | 21585.30 (7915.479) | 9653.80 (4245.794)
  Last Dose: EP-038725 | 8944.82 (4528.012) | 2588.19 (1379.765)
  Last Dose: EP-039082: number analyzed (Participants) | 39 | 22
  Last Dose: EP-039082 | 48.21 (26.600) | 7.31 (10.464)

29. Secondary Outcome: Number of Participants With Adverse Events (AEs) up to Discharge
Description: An AE was defined as any untoward medical occurrence in clinical study participants administered a pharmaceutical (investigational or non-investigation) product. An AE does not necessarily have a causal relationship with the study intervention. A serious AE (SAE) was defined as any untoward medical occurrence that, at any dose:
  * Resulted in death
  * Was life threatening
  * Required inpatient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent disability/incapacity
  * Was a congenital anomaly/birth defect
  * Was an important medical event
Time Frame: Day -2 to Day 12
Population: Safety Analysis Set (Treated Participants): All participants having received challenge virus and IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 47 | 47 | 47
Participants
  Any AE | 13 | 15 | 15
  Any SAE | 0 | 0 | 0

30. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An AE was defined as any untoward medical occurrence in clinical study participants administered a pharmaceutical (investigational or non-investigation) product. An AE does not necessarily have a causal relationship with the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose:
  * Resulted in death
  * Was life threatening
  * Required inpatient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent disability/incapacity
  * Was a congenital anomaly/birth defect
  * Was an important medical event
Time Frame: Day 1 to Day 28
Population: Safety Analysis Set (Treated Participants): All participants having received challenge virus and IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo
Number analyzed (Participants) | 47 | 47 | 47
Participants
  Any TEAEs | 11 | 14 | 13
  Any Treatment-emergent SAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: Day -2 to Day 28; all adverse events: Day -2 to Day 28
Description: All-cause mortality: Safety Analysis Set - All participants having received challenge virus, regardless of whether they received IMP or not; Adverse events: Safety Analysis Set (Treated Participants) - All participants having received challenge virus and IMP
Arm/Group | EDP-323 High Dose | EDP-323 Low Dose | Placebo | Enrolled But Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47 | 0/47 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/47 | 0/0
Other Adverse Events (participants affected / at risk) | 13/47 | 15/47 | 15/47 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EDP-323 High Dose (N=47) | EDP-323 Low Dose (N=47) | Placebo (N=47) | Enrolled But Not Randomized (N=0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diagnostic procedure (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vessel puncture site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival hyperemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT06170242/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT06170242/SAP_001.pdf